CLINICAL TRIAL: NCT00762944
Title: Survivibility of the Total Temporomandibular Joint Replacement System
Brief Title: Total Temporomandibular Joint Replacement System Post Approval Study
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: BMET WL 01
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Arthroplasty
Keywords: Patients requiring total joint reconstruction due to:; Arthritis (osteo-, rheumatoid, traumatic) malignancy; Ankylosis functional deformity; Avascular necrosis revisions; Benign neoplasms fracture; Multiple operated joints
MeSH Terms: conditions — Arthritis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Biomet TMJ Replacement System: All patients required total reconstruction of the temporomandibular joint (unilateral or billateral)
  Interventions: Device: Biomet TMJ Replacement System

INTERVENTIONS:
Device: Biomet TMJ Replacement System — Total replacement of the temporomandibular joint with a Biomet TMJ Replacement System
  Other Names: TMJ alloplastic reconstruction

SUMMARY:
Post-Approval Study (PMA CoA) in Order to Obtain Additional Long Term Safety and Effectiveness Data [PMA P020016]

DETAILED DESCRIPTION:
An additional three-year follow-up data will be collected on subjects previously enrolled in the PMA study, who had not completed follow-up prior to the PMA approval [PMA P020016].

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring total joint reconstruction due to:

   Arthritis (osteoarthritis, rheumatoid, traumatic) malignancy Ankylosis functional deformity Avascular necrosis revisions Benign neoplasms fracture Multiple operated joints
2. Patients who are skeletally mature.
3. Patients must have at least one of the following criteria for surgical TMJ treatment.

   1. Presence of considerable pain and/or limited function in the joint area.
   2. Clinical and imaging evidence consistent with anatomic joint pathology
   3. Previous failure of non-surgical treatment/therapy or a failed implant.
   4. High probability of patient improvement by surgical treatment.
4. Patients must be able to return for follow-up examinations.
5. Patients without serious compromising general medical conditions.

Exclusion Criteria:

1. Patients with active infection.
2. Patient conditions where there is insufficient quantity or quality of bone to support the device
3. Patients with perforations in the mandibular fossa and/or bony deficiencies in the articular eminence compromising support for the artificial fossa component.
4. Patients with mandibular and/or zygomatic arch screw holes compromising component fixation
5. Patients requiring partial joint reconstruction or other TMJ procedures not listed as an indication.
6. Patients who are NOT skeletally mature.
7. Patients who are incapable or unwilling to follow postoperative care instructions.
8. Patients who are unable to return for follow-up examinations.
9. Patients with severe hyper-functional habits
10. Patients on chronic steroid therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received TMJ systems from the IDE study
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2005-09-21 (Actual); Primary Completion 2008-08-25 (Actual); Study Completion 2008-09-21 (Actual)

PRIMARY OUTCOMES:
Time to Revision | 3 years
  Time from surgical alloplastic reconstruction of the TMJ to revision surgery (Re-operation or removal)

SECONDARY OUTCOMES:
jaw pain intensity (VAS score) | 1 year, 1.5 years
  Pain level is recored in a 10 cm line according the intensity of pain, where zero on the far left represents "no pain" and 10 on the far right, represent the maximum level of pain experienced
Interference with eating | 1 year, 1.5 years
  Interference of eating is recored in a 10 cm line according the intensity of the interference with eating, where zero on the far left represents "no interference with eating" and 10 on the far right, represent the maximum level of interference with eating experienced
Maximun Incisal Opening | 1 year, 1.5 years
  Maximum Incisal Opening (MIO) is the distance measured in millimeters (mm) from the incisal edge of the maxillary central incisors to the incisal edge of the mandibular central incisors at the midline with the mouth wide open.
Patient Satisfaction | 6 months, 1 year, 1.5 years, and 3 years
  Patient satisfaction is the level of comfort with the TMJ reconstruction that a given patient experiences. It is expressed as "very satisfied", "satisfied", "dissatisfied" or "failure"

CONTACTS AND LOCATIONS:
Overall Officials: Oscar A Gonzalez, MD, DNP, Study Chair — Zimmer Biomet
Locations (4):
- United States (4):
  - Riley Hospital, Indianapolis, Indiana
  - Jeffrey S. Topf, D.D.S., West Bloomfield, Michigan
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas,Southwestern Medical School, Dallas, Texas